CLINICAL TRIAL: NCT06284330
Title: CHARGE: CHOICE ARCHITECTURE IN GENETIC TESTING
Brief Title: CHARGE Study: CHoice ARchitecture Genetic tEsting
Acronym: CHARGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sukh Makhnoon, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU-2023-0881
Record Dates: First submitted 2024-02-01; First posted 2024-02-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Cancer
Keywords: cascade genetic testing; hybrid type I; feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care cascade testing (No Intervention): Standard of care cascade genetic testing
- Choice architecture cascade testing (Experimental): Direct mailed genetic testing kit to probands' relatives.
  Interventions: Other: Enhanced cascade testing

INTERVENTIONS:
Other: Enhanced cascade testing — Direct mailed at-home genetic testing kit to probands' relatives.
  Arms: Choice architecture cascade testing

SUMMARY:
CHARGE is a hybrid type I feasibility study to compare a choice architecture intervention for cascade genetic testing to usual care.

DETAILED DESCRIPTION:
CHARGE study contains two arms: Arm 1) Usual care, comprising of standard genetic counseling and education to probands regarding cascade testing; and Arm 2) Direct mailing of a home genetic testing kit to probands' at-risk relatives that can be returned directly to a commercial genetic testing laboratory, including educational information on the importance and cost of cascade testing

ELIGIBILITY:
Proband Inclusion Criteria:

* Have a newly reported pathogenic or likely pathogenic variant in one or more of the following genes: APC, ATM, BRCA1, BRCA2, CDH1, CHEK2, PALB2, MLH1, MSH2, MSH6, PMS2, PTEN, TP53
* 18 years of age or older
* English fluency
* Have at least 1 adult living genetically related relative who resides in Texas

Proband Exclusion Criteria:

* Referred for genetic testing by a relative with a pathogenic variant
* Unwilling to be randomized to a study arm

Relative Inclusion Criteria:

* 18 years of age or older
* English fluency
* Residing in Texas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of cascade genetic testing | 3-6 months
  Proportion of at-risk relatives who undergo testing

SECONDARY OUTCOMES:
Change in probands' family communication about genetic test results as measured by Proband survey | Baseline and 4-7 months
  Frequency and content of family communication will be measured by Proband survey (result sharing, reasons for sharing and not sharing)
Proband's and relative's satisfaction with decision about participating in study measured at approximately 4- 7 months | Approx. 4-7 months
  Probands' and relative's satisfaction with decision about participating in study will be measured at approximately 4- 7 months using surveys (intervention arm). This is measured using the satisfaction with decision scale.
Family functioning as reported by probands and relatives measured by Cancer Family Impact Scale | 4-7 months
  Relatives' and probands' family functioning will be measured by a survey that includes the adapted Cancer Family Impact Scale. Participants responses to the 18 items of CFIS on a 5-point Likert scale are summed for scoring. Higher summed scores indicated a greater communication and flow of about cancer information within family and therefore better family functioning.
Proband's reaction to intervention materials as measured by proband survey. | 4-7 months
  Proband survey will include adapted versions of usability questions, commonly used in usability tests of eHealth tools that assess satisfaction, liking, ease of use, and preference. Possible scores range from 0-5 where lower score indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sukh Makhnoon, PhD, MS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makhnoon S, Getchell G, Rodriguez Y, Pena L, Rodriguez J, Ibidapo T, Henrikson NB, Lee M, Wu S, Pirzadeh-Miller S. Choice architecture in cascade genetic testing (CHARGE study) for hereditary cancer: Design of a hybrid type I randomized feasibility trial. Contemp Clin Trials. 2025 Aug;155:107979. doi: 10.1016/j.cct.2025.107979. Epub 2025 Jun 5. PMID 40482962